CLINICAL TRIAL: NCT03790618
Title: Effect of Stimulant Drugs on Social Perception
Acronym: ESP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB15-780
Record Dates: First submitted 2018-11-30; First posted 2018-12-31 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Healthy; MDMA ('Ecstasy')
MeSH Terms: interventions — Methamphetamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects will attend one session during which they will receive a placebo capsule.
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: methamphetamine
- Low dose MDMA (Experimental): Subjects will attend one session during which they will receive 0.75mg/kg MDMA.
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: methamphetamine
- High dose MDMA (Experimental): Subjects will attend one session during which they will receive 1.5mg/kg MDMA.
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: methamphetamine
- Methamphetamine (Experimental): Subjects will attend one session during which they will receive 20mg methamphetamine.
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: methamphetamine

INTERVENTIONS:
Drug: 3,4-Methylenedioxymethamphetamine — Participants will be given 0.75mg/kg of 1.5mg/kg MDMA
Drug: methamphetamine — Please see above.

SUMMARY:
The study will improve our understanding of the "prosocial" effects of ± 3,4-Methylenedioxymethamphetamine (MDMA), relative to a prototypical stimulant, methamphetamine (MA). The investigators seek to characterize the "uniquely social" effects of MDMA.

ELIGIBILITY:
Inclusion Criteria:

* High school degree
* English fluency
* Healthy
* Has used MDMA

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Any medical or psychiatry condition

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bershad AK, Hsu DT, de Wit H. MDMA enhances positive affective responses to social feedback. J Psychopharmacol. 2024 Mar;38(3):297-304. doi: 10.1177/02698811231224153. Epub 2024 Jan 27. PMID 38279662

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Low Dose MDMA | High Dose MDMA | Methamphetamine
Started | 9 | 9 | 9 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose MDMA | High Dose MDMA | Methamphetamine | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 9 | 9 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 5 | 5 | 20
  Male | 4 | 4 | 4 | 4 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 2 | 8
  White | 5 | 5 | 5 | 5 | 20
  More than one race | 1 | 1 | 1 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 9 | 36
Education - High School Education [Count of Participants; unit: Participants] | 9 | 9 | 9 | 9 | 36

OUTCOME MEASURES:

1. Primary Outcome: Responses to Affective Touch
Description: Participants will complete an affective touch task during which time they will rate pleasantness of touch on a likert scale of 1-7, with higher scores indicating greater ratings of pleasantness
Time Frame: End of study (time 0 and approximately six weeks later)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose MDMA | High Dose MDMA | Methamphetamine
Number analyzed (Participants) | 9 | 9 | 9 | 9
units on a scale | -1.24 (3.22) | 0.12 (3.14) | 0.19 (2.25) | 0.25 (2.68)

ADVERSE EVENTS:
Time Frame: period of time was until completion which was six weeks on average.
Arm/Group | Placebo | Low Dose MDMA | High Dose MDMA | Methamphetamine
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT03790618/Prot_SAP_000.pdf